CLINICAL TRIAL: NCT06011278
Title: The Effect of Community-Provided Psychosocial Support Videos on Disease Attitudes and Symptoms of Pediatric Oncology Patients
Brief Title: The Effect of Community-Provided Psychosocial Support Videos on Disease Attitudes and Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Teaching Assisstant, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EysanU
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Assignment to the experimental and control groups will be made by an independent statistician to avoid bias and ensure confidentiality. Thus, selection bias will be controlled by making random assignment and hiding the randomization.
  In the study, participant and researcher will not be blinded. Blinding will not be possible because the researcher follows the participants and parents on a daily basis and is aware of the intervention. The data will be coded as 'A' and 'B' by the researcher and transferred to the computer. It is recommended that all stages of randomized controlled trials be conducted according to the Consolidated Standards of Reporting Trials (CONSORT). In this context, the study will be conducted on the basis of the CONSORT 2017 (Updated Guidelines for Reporting Randomized Parallel Group Studies) guideline during the randomization stages of this study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-supported videos (Experimental): Community-supported videos will be sent to the children in the experimental group once a week for a month. At the end of four weeks, the "Chıld Attıtude Toward Illness Scale" and the "Memorial Symptom Assessment Scale" will be administered to the children again.
  Interventions: Other: Community Supported Videos
- Standard care (No Intervention): Children in the control group will receive the standard care of the pediatric oncology clinic.At the end of four weeks, the "Chıld Attıtude Toward Illness Scale" and the "Memorial Symptom Assessment Scale" will be administered to the children again.

INTERVENTIONS:
Other: Community Supported Videos — Volunteers will be asked to create a maximum of three minutes of content that will psychosocially strengthen and motivate pediatric oncology patients. In the videos, information will be given about not using words such as cancer/oncology/tumor and not including private and personal information. Videos will be created in such a way that they can be edited, merged or deleted accordingly. The applications of volunteer individuals will be made through social media (Instagram), the collection of these videos will be followed in accordance with the voluntary consent forms, and the volunteers will be informed in detail about the use of visual and verbal data.
  Children will be sent videos featuring different volunteers each week. The content of the videos will be controlled by the child clinical psychologist and researchers. Inappropriate videos will not be included in the research.
  Arms: Community-supported videos

SUMMARY:
The effects of psychosocial support on the disease process have been studied with many different groups and diseases, and even the psychosocial support needed by the family of the child with a chronic disease has been the subject of research, but studies focusing directly on the needs of the child have been very limited. Although it is seen in the existing literature that studies such as art and play therapy or educational programs have been carried out to improve the attitudes of pediatric oncology patients towards their own diseases, no study has been found that investigated the effects of social/social support in pediatric oncology patients. In order to contribute to this limitation in the literature, this study aimed to examine the effects of community-provided psychosocial support videos on the attitudes and symptoms of pediatric oncology patients.

DETAILED DESCRIPTION:
Cancer can affect every individual regardless of age and gender, causing individuals to experience a situation they were not used to before. People may not be able to apply the coping mechanisms they know or they may not find enough coping strength in themselves. This situation can cause individuals to experience emotions such as fear, anxiety and stress. At the beginning of the periods when the diagnosis of cancer is particularly difficult to cope with, comes the period of adolescence and adolescence, which covers the age range of 10-18, in which we plan to conduct the research.

During this period, relationships with people other than parents gained importance; the interest is on peers and non-peer social relationships; It is a developmental period in which there are sudden fluctuations in emotions, especially due to physical changes, and in which he is more inclined to isolate himself from the social environment. They need external approval and encouragement in the changes that occur with their physical and mental developments. Even in healthy children, the lack of this approval and social support may result in a negative development; Pediatric oncology patients are more vulnerable due to the side effects of the disease and treatment process or the physical and psychological effects it causes. For children whose psychosocial development continues, being diagnosed with cancer causes an additional difficulty in their developmental processes. Because children have less or inadequate coping mechanisms than the average adult during this period; This may make it difficult to accept the disease due to the negative effects of diagnosis and treatment.

This period, which is considered more vulnerable to trauma, makes the situation more complicated and tiring for a pediatric oncology patient compared to an adult cancer patient. For this reason, it is very important to control and manage the attitudes of patients towards their own diseases. Minimizing psychosocial problems in order to get the best benefit from the treatment process will also increase the patient's efficiency from the treatment. In this study, it is aimed to evaluate the effect of the psychosocial support videos provided by the community to pediatric oncology patients aged 10-18 on the children's attitudes towards their own disease and treatment-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* In the 10-18 age group,
* Newly diagnosed with cancer (maximum three months ago),
* Ongoing active treatment,
* Speaking in Turkish,
* Having no visual, auditory, and mental problems,
* Knowing the diagnosis,
* Children who volunteer to participate in the research and their parents will be included.

Exclusion Criteria:

* The hospitalization period is less than 4 weeks,
* Neutropenic children,
* In the terminal period,
* With intense pain expression,
* Being under any sedative/anticonvulsant/analgesic effect,
* Children and their parents who apply to the hospital with a life-threatening illness/condition will not be included.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-08 (Estimated); Study Completion 2023-09-11 (Estimated)

PRIMARY OUTCOMES:
Chıld Attıtude Toward Illness Scale | Three week
  It was developed to measure the attitudes of children with chronic diseases towards their own diseases. During the evaluation, the scores obtained from 13 items are added and divided into 13 or according to the number of items.The total score range is 1 to 5. A score of 1 and 2 indicates negative attitude, 3 indicates neutral attitude, and 4 and 5 indicates positive attitude.

SECONDARY OUTCOMES:
Memorial Symptom Assessment Scale | Three week
  The Memorial Symptom Assessment Scale is developed to determine the symptoms experienced in the last week of children aged 10-18 years who are followed up with the diagnosis of cancer. your scale; It has three sub-dimensions: physical, psychological and general condition index. The Turkish validity and reliability of the scale was done by Atay et al.The lowest score is 30 and the highest score is 120. A high score indicates that the symptom is high in frequency, severity, and distress for the child.

CONTACTS AND LOCATIONS:
Overall Officials: Eyşan Umaç, MsC, Study Chair — Koç University
Locations (1):
- Koc University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No